CLINICAL TRIAL: NCT02454647
Title: Induction Chemotherapy, Chemo-radiotherapy and Surgery in Locally Advanced Gastric Cancer Patients: Long Term Results From a Single Institution.
Brief Title: Induction Chemotherapy, Chemoradiotherapy and Surgery in Locally Advanced Gastric Cancer Patients
Status: Completed | Type: Observational
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Other Study IDs: GC-PKPDGN
Record Dates: First submitted 2015-05-22; First posted 2015-05-27 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Gastric Cancer; Adenocarcinoma; Effects of Chemotherapy; Surgery; Gastrointestinal Neoplasms
Keywords: Radiotherapy; Neoadjuvant therapy; Induction chemotherapy; Concurrent chemoradiotherapy; Preoperative factors; Dynamic factors; Prognostic Factor
MeSH Terms: conditions — Stomach Neoplasms; Adenocarcinoma; Gastrointestinal Neoplasms | interventions — Induction Chemotherapy; Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Surgical specimen with potential for extraction of DNA.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Induction chemotherapy
Radiation: Radiotherapy with concurrent chemotherapy
Procedure: Salvage surgery

SUMMARY:
The aim of this study is to evaluate the efficacy of a neoadjuvant approach in patients with locally advanced gastric cancer and the identification of prognostic factors.

DETAILED DESCRIPTION:
Patients with locally advanced gastric cancer (T3-4 and/or N+) are included. Initially, patients are diagnosed by computerized tomography scan and endoscopic ultrasound.

The neoadjuvant strategy consists of 3-4 cycles of induction chemotherapy followed by concurrent chemoradiotherapy. Chemoradiotherapy comprises weekly chemotherapy concurrently with daily external beam radiotherapy up to 45 Gy). Surgery is scheduled 4 to 6 weeks after the end of CRT. Pathological response is graded according to the Becker criteria. Statistical analysis is performed IBM SPSS v20.

Estimate whether R0 resection rate, pathological response degree, patterns of recurrence and long-term outcomes may be initially predicted by dynamic prognostic factors as tumor size, neutrophil lymphocyte ratio (NLR) and platelet lymphocyte ratio (PLR)

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the stomach
* Age ≥18 years old
* Performance Status- Eastern Cooperative Oncology Group (ECOG) 0-1
* Body mass index ≥ 18
* No prior chemotherapy or chemoradiotherapy
* TNM stage of T3-T4 and/or positive regional lymph nodes (N+) by endoscopic ultrasound or computed tomography (CT)
* No evidence of metastasis (M0)
* Adequate hematological, liver and renal functions (ALT and AST≤2.5 UNL, total bilirubin ≤1.5 UNL, and serum creatinine ≤1.5 UNL)

Exclusion Criteria:

* Patients with previous (less than 10 years) or current history of malignant neoplasms, except for curatively treated
* Patients with evidence of severe or uncontrolled systemic disease
* Medically unfit for chemotherapy
* Tumors involving the esophageal junction, comprising siewert I to III

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with locally advanced adenocarcinoma of the stomach treated with a neoadjuvant protocol consisting of induction chemotherapy (ICT), chemoradiotherapy (CRT)and salvage surgery. Patients must have a medically fit condition to complete the protocol.
  Initial staging comprises a thoracic and abdominal computerised tomography scan, endoscopic ultrasound endoscopy (EUS), biopsy and blood test including blood cell count, hepatic and renal function.
  Radiological and endoscopic evaluations are performed at baseline and at the completion of ICT and CRT.
  Blood tests are acquired at baseline, before each chemotherapy course and concurrently with evaluations. Blood tests are also obtained during follow-up and at the time progression.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2013-09; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Overall Survival | From date of treatment until death, assessed up to 10 years
  Overall was defined as the period from diagnosis until death (from any cause).
Identification of prognostic factors for overall survival | From date of treatment until death, assessed up to 10 years
  Overall was defined as the period from diagnosis until death (from any cause). Correlation between survival and baseline, clinical and treatment characteristics from patients
Disease-free survival | From date of diagnosis until progression or death, assessed up to 10 years
  Disease-free survival was defined as the time from diagnosis to the first date of local or distant cancer.
R0 resection rate | Week 24 to 28
  The R0 resection rate in the patients treated with the neoadjuvant protocol. R0 is defined as a microscopically margin-negative resection, in which no gross or microscopic tumor remains in the primary tumor bed.

SECONDARY OUTCOMES:
Pathological response | Week 24 to 28
  Specimen analysis according to TNM classification. Pathological complete response is defined as no invasive cancer cells in the surgical specimen.
Patterns of treatment failure | From date of diagnosis until treatment failure, assessed up to 10 years
  Type of recurrence: local, regional and/or distant.
Adverse events are assessed according to CTC criteria v 4.0 | Week 1 to 20
  Safety and tolerability during the neoadjuvant protocol.

CONTACTS AND LOCATIONS:
Overall Officials: javier Rodriguez Rodriguez, MD, PhD, Principal Investigator — CUN
Locations (1):
- Clinica Universidad de Navarra, Pamplona, Navarre, Spain